CLINICAL TRIAL: NCT00418379
Title: A Randomised, Double-blind, Placebo-controlled, Multi-national, Multi-centre, Phase III Study to Assess the Long Term Efficacy, Carry-over Effect and Safety of Two Dosing Regimens of 300 IR Sublingual Immunotherapy (SLIT) Administered as Allergen-based Tablets Once Daily to Patients Suffering From Grass Pollen Rhinoconjunctivitis
Brief Title: Phase III Study to Assess the Long Term Efficacy, Carry-over Effect and Safety of 300 IR Sublingual Immunotherapy Tablets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VO53.06
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Allergy
Keywords: Sublingual immunotherapy; Grass pollen tablet; Allergic rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 300 IR (4M) (Experimental): 300 IR grass pollen allergen extract tablet, treatment starting 4 months before the pollen season
  Interventions: Drug: 300 IR (4M)
- 300 IR (2M) (Experimental): 300 IR grass pollen allergen extract tablet, treatment starting 2 months before the pollen season
  Interventions: Drug: 300 IR (2M)
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 300 IR (4M) — 300 IR grass pollen allergen extract tablet starting 4 months before the pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR (4M)
Drug: 300 IR (2M) — 300 IR grass pollen allergen extract tablet starting 2 months before the pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR (2M)
Drug: Placebo — Placebo tablet
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
A phase III study to evaluate Long term efficacy , carry-over effect and safety of 300 IR sublingual Immunotherapy (SLIT) tablets in adults patients suffering from grass pollen rhinoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 to 50 years
* Grass pollen-related allergic rhinoconjunctivitis for at least the last two pollen seasons
* Positive SPT and specific IgE values of at least Class 2 for grass pollen allergens
* A score of greater than or equal to 12 out of a possible 18 on the Retrospective Rhinoconjunctivitis Total Symptom Score (RRTSS)

Exclusion Criteria:

* Patients with symptoms of rhinoconjunctivitis during the grass pollen season due to sensitisation to allergens other than grass pollen must not be included. Patients must be asymptomatic to all other allergens during the grass pollen season. Patients who have allergic rhinitis due to perennial allergen may not be included.
* Asthma requiring treatment other than beta-2 inhaled agonists.
* Patients who have received any desensitisation treatment for grass pollen or with any other allergen within the previous 5 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 633 (Actual)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain DIDIER, MD, Pr, Principal Investigator — Hôpital Rangueil-Larrey, Toulouse, France
Locations (1):
- DIDIER, Toulouse, France

REFERENCES:
- [Result] Didier A, Worm M, Horak F, Sussman G, de Beaumont O, Le Gall M, Melac M, Malling HJ. Sustained 3-year efficacy of pre- and coseasonal 5-grass-pollen sublingual immunotherapy tablets in patients with grass pollen-induced rhinoconjunctivitis. J Allergy Clin Immunol. 2011 Sep;128(3):559-66. doi: 10.1016/j.jaci.2011.06.022. Epub 2011 Jul 29. PMID 21802126
- [Result] Didier A, Malling HJ, Worm M, Horak F, Sussman G, Melac M, Soulie S, Zeldin RK. Post-treatment efficacy of discontinuous treatment with 300IR 5-grass pollen sublingual tablet in adults with grass pollen-induced allergic rhinoconjunctivitis. Clin Exp Allergy. 2013 May;43(5):568-77. doi: 10.1111/cea.12100. PMID 23600548
- [Derived] Didier A, Malling HJ, Worm M, Horak F, Sussman GL. Prolonged efficacy of the 300IR 5-grass pollen tablet up to 2 years after treatment cessation, as measured by a recommended daily combined score. Clin Transl Allergy. 2015 May 22;5:12. doi: 10.1186/s13601-015-0057-8. eCollection 2015. PMID 26097680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 08 DEC 2006, Last Patient Last Visit 07 SEP 2011
Period: Year 1
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Started | 207 | 207 | 219
Completed | 189 | 179 | 204
Not Completed | 18 | 28 | 15
Not completed — Adverse Event | 9 | 15 | 3
Not completed — Withdrawal by Subject | 7 | 8 | 5
Not completed — Any other reason not above-mentioned | 2 | 5 | 7
Period: Year 2
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Started | 167 (22 patients withdrew between Year 1 and Year 2 treatment periods.) | 159 (20 patients withdrew between Year 1 and Year 2 treatment periods.) | 182 (22 patients withdrew between Year 1 and Year 2 treatment periods.)
Completed | 159 | 155 | 172
Not Completed | 8 | 4 | 10
Not completed — Adverse Event | 5 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Any other reason not above-mentioned | 2 | 1 | 6
Period: Year 3
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Started | 151 (8 patients withdrew between Year 2 and Year 3 treatment periods.) | 148 (7 patients withdrew between Year 2 and Year 3 treatment periods.) | 166 (6 patients withdrew between Year 2 and Year 3 treatment periods.)
Completed | 148 | 146 | 163
Not Completed | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Any other reason not above-mentioned | 2 | 1 | 1
Period: Year 4
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Started | 145 (3 patients withdrew between Year 3 and Year 4 study periods.) | 141 (5 patients withdrew between Year 3 and Year 4 study periods.) | 156 (7 patients withdrew between Year 3 and Year 4 study periods.)
Completed | 142 | 136 | 154
Not Completed | 3 | 5 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Any other reason not above-mentioned | 1 | 1 | 0
Period: Year 5
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Started | 128 (14 patients withdrew between Year 4 and Year 5 study periods.) | 120 (16 patients withdrew between Year 4 and Year 5 study periods.) | 134 (20 patients withdrew between Year 4 and Year 5 study periods.)
Completed | 126 | 115 | 131
Not Completed | 2 | 5 | 3
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Any other reason not above-mentioned | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set Year 1 (FASY1). FASY1 included all patients who received at least one dose of the investigational product and had at least one Adjusted Symptom Score (ASS) during the pollen period while on treatment during the Year 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo | Total
Number analyzed (Participants) | 188 | 188 | 205 | 581
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (8.25) | 30.4 (7.57) | 30.2 (8.56) | 30.5 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 77 | 83 | 226
  Male | 122 | 111 | 122 | 355

OUTCOME MEASURES:

1. Primary Outcome: Average Adjusted Symptom Score (AAdSS)
Description: The Adjusted Symptom Score (AdSS) is a subject-specific symptom score which is adjusted for rescue medication use.
  Participants assessed daily, during the Year 3 pollen period while on treatment, 6 rhinoconjunctivitis symptoms (sneezing, rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes) each symptom is scored as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms. The sum of the 6 symptoms is the Rhinoconjunctivitis Total Symptom Score (RTSS) (range 0-18). If the subject took rescue medication on a given day, the AdSS equals the RTSS of that day or the AdSS of the day before, whichever is higher. This adjustment applies to the day of rescue medication use and the following day. Like the RTSS, the AdSS ranges from 0 to 18. The lower the score, the better the outcome.
Time Frame: Pollen period (average of 33.8 days) of Year 3
Population: Full Analysis Set Year 3 (FASY3). FASY3 included all patients who received at least one dose of the investigational product and had at least one Adjusted Symptom Score (AdSS) during the pollen period while on treatment during the Year 3.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (range: 0 to 18)
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Number analyzed (Participants) | 149 | 147 | 165
Units on a scale (range: 0 to 18) | 3.39 (0.357) | 3.25 (0.369) | 5.21 (0.348)
Statistical Analysis 1: Comparison: 300 IR (4M) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: 300 IR (2M) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Over 3 years during the treatment periods .
Description: TEAEs were defined as any AE which started on or after the administration of the investigational product (IP) in the corresponding treatment period up to 30 days after the last administration of the IP (inclusive) for the corresponding period.
  Note: Serious Adverse Events and Other Adverse Events are described in the Results Publications.
Arm/Group | 300 IR (4M) | 300 IR (2M) | Placebo
Serious Adverse Events (participants affected / at risk) | 9/207 | 7/207 | 6/219
Other Adverse Events (participants affected / at risk) | 179/207 | 167/207 | 170/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 300 IR (4M) (N=207) | 300 IR (2M) (N=207) | Placebo (N=219)
APPENDICITIS (Infections and infestations) | 1 | 0 | 0
DIARRHOEA (Infections and infestations) | 1 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 0 | 1
GENITAL INFECTION (Infections and infestations) | 1 | 0 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 1 | 0
BENIGN NEOPLASM OF CERVIX UTERI (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
TESTICULAR GERM CELL TUMOUR MIXED STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
FAMILIAL MEDITERRANEAN FEVER (Congenital, familial and genetic disorders) | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0/167 | 0/159 | 1/182
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1/167 | 0/159 | 0/182
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0/167 | 1/159 | 0/182
ABORTION INDUCED (Surgical and medical procedures) | 0/167 | 1/159 | 0/182
EYE INJURY (Injury, poisoning and procedural complications) | 1/151 | 0/148 | 0/166
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0/151 | 1/148 | 0/166
GASTROENTERITIS (Infections and infestations) | 0/151 | 0/148 | 1/166
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0/151 | 1/148 | 0/166
RENAL COLIC (Renal and urinary disorders) | 0/151 | 0/148 | 1/166
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0/151 | 0/148 | 1/166
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (4M) (N=207) | 300 IR (2M) (N=207) | Placebo (N=219)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 70 | 60 | 20
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 36 | 35 | 41
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 35 | 33 | 38
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 27 | 28 | 37
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 26 | 26 | 33
COUGH (Respiratory, thoracic and mediastinal disorders) | 31 | 33 | 34
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 18 | 19 | 13
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 12 | 21 | 14
ORAL PRURITUS (Gastrointestinal disorders) | 107 | 89 | 32
OEDEMA MOUTH (Gastrointestinal disorders) | 26 | 17 | 3
DYSPEPSIA (Gastrointestinal disorders) | 13 | 10 | 1
EYE PRURITUS (Eye disorders) | 30 | 33 | 39
LACRIMATION INCREASED (Eye disorders) | 16 | 22 | 28
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 11 | 14 | 21
CONJUNCTIVITIS (Eye disorders) | 14 | 17 | 13
NASOPHARYNGITIS (Infections and infestations) | 42 | 26 | 46
RHINITIS (Infections and infestations) | 16 | 16 | 13
HEADACHE (Nervous system disorders) | 23 | 28 | 46
EAR PRURITUS (Ear and labyrinth disorders) | 32 | 15 | 5
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 14 | 12 | 17
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 2
ORAL DISCOMFORT (Gastrointestinal disorders) | 13 | 12 | 3
GLOSSODYNIA (Gastrointestinal disorders) | 11 | 8 | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 11 | 6 | 1
PHARYNGITIS (Infections and infestations) | 10 | 16 | 19
INFLUENZA (Infections and infestations) | 12 | 7 | 13
SEASONAL ALLERGY (Immune system disorders) | 11 | 10 | 15
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 7 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No